CLINICAL TRIAL: NCT04247321
Title: Non-invasive Near-infrared Spectroscopy (NIRS) Versus Invasive Licox Intracranial Pressure Monitoring in Neurocritical Care
Brief Title: Non-invasive Near-infrared Spectroscopy (NIRS) Versus Invasive Licox Intracranial Pressure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: • Withdrawn: Study halted prematurely, prior to enrollment of first participant
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alejandro Rabinstein, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 19-008406
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Subjects with acute brain injury (Experimental): Subjects requiring placement of a Licox Brain Tissue Oxygen device for their clinical care will also have Near-infrared spectroscopy (NIRS) monitoring system placed
  Interventions: Device: Licox® Brain Tissue Oxygen Monitoring System; Device: Near-infrared spectroscopy (NIRS)

INTERVENTIONS:
Device: Licox® Brain Tissue Oxygen Monitoring System — Invasive brain tissue oxygenation monitoring
Device: Near-infrared spectroscopy (NIRS) — Non-invasive approach to monitoring brain tissue oxygenation which uses two wavelengths of near infrared light and takes measurements of the ratio of oxyhemoglobin to total hemoglobin

SUMMARY:
Researchers are trying to assess how accurately and safely NIRS non-invasive monitoring can detect changes in intracranial pressure to determine if this noninvasive device can be used instead of invasive monitoring with Licox in the future.

ELIGIBILITY:
Inclusion:

* Subjects with acute brain injury who are age ≥ 18
* Glasgow coma scale score (GCS) ≤ 8
* Neuroimaging concerning for ICP crises, or have active ICP treatment
* Have Licox Brain Tissue Oxygen monitor placed as standard of care treatment

Exclusion:

* CNS infection
* Bleeding diathesis or thrombocytopenia < 50,000 platelets
* Subjects with subdural hematomas who have had surgical decompression and bone flap removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between changes in Licox and NIRS oxygenation measurements | 3 to 5 days of the monitoring duration
  Licox measures oxygenation in terms of partial pressure (PtO2) and NIRS measures it in terms of saturation (rSO2). The changes in PtO2 versus the changes in rSO2 will be compared for equivalence.

SECONDARY OUTCOMES:
Correlation between changes in pressure reactivity index and Licox versus NIRS | 3 to 5 days of the monitoring duration
  The pressure reactivity index (PRx) is derived using ICM+ software; the PRx is a correlation coefficient ranging from -1 to +1; PRx > 0 indicates poor autoregulation. We will investigate if PRx correlates with changes in rSO2 as measured by NIRS (if changes in autoregulation correspond with changes in oxygenation).

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro A Rabinstein, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials